CLINICAL TRIAL: NCT00550238
Title: A Multi-Center, Open-Label Extension Study to Examine the Safety and Tolerability of ACP-103 in the Treatment of Psychosis in Parkinson's Disease
Brief Title: A Study of the Safety and Tolerability of Pimavanserin (ACP-103) in Patients With Parkinson's Disease Psychosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-103-015
Record Dates: First submitted 2007-10-26; First posted 2007-10-29 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-05

CONDITIONS: Parkinson's Disease Psychosis
Keywords: Parkinson's Disease Psychosis
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pimavanserin tartrate (ACP-103) (Experimental): Tablets taken once daily by mouth for as long as ACP-103 is considered to be tolerated and beneficial to subjects
  Interventions: Drug: Pimavanserin tartrate (ACP-103)

INTERVENTIONS:
Drug: Pimavanserin tartrate (ACP-103) — Tablets taken once daily by mouth for as long as ACP-103 is considered to be tolerated and beneficial to subjects

SUMMARY:
To assess the long-term safety and tolerability of ACP-103 in subjects with Parkinson's disease psychosis.

DETAILED DESCRIPTION:
This study did not have a fixed duration, and the duration of individual subject participation was determined based on investigator assessment of subject tolerability and continued benefit until such time as either the drug was commercially available in the US, or an alternate treatment extension was available in non-US regions. For this reason, no subjects, therefore, were considered to have "completed" the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject has completed the treatment period of a previous blinded study of pimavanserin
* The subject is willing and able to provide consent
* Caregiver is willing and able to accompany the subject to all visits

Exclusion Criteria:

* Subject has current evidence of a serious and or unstable cardiovascular, respiratory, gastrointestinal, renal, hematologic or other medical disorder
* Subject is judged by the Investigator to be inappropriate for the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2007-07; Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (130):
- United States (83):
  - Gilbert, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Berkeley, California
  - Carson, California
  - Fountain Valley, California
  - Fresno, California
  - Irvine, California
  - La Habra, California
  - La Jolla, California
  - Laguna Hills, California
  - Loma Linda, California
  - Oxnard, California
  - Pasadena, California
  - Reseda, California
  - Sunnyvale, California
  - Ventura, California
  - Englewood, Colorado
  - Danbury, Connecticut
  - Fairfield, Connecticut
  - Farmington, Connecticut
  - Boca Raton, Florida
  - Bradenton, Florida
  - Deerfield Beach, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Naples, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Panama City, Florida
  - Pompano Beach, Florida
  - Port Charlotte, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Decatur, Georgia
  - Glenview, Illinois
  - Springfield, Illinois
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Scarborough, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Clinton Township, Michigan
  - Detroit, Michigan
  - East Lansing, Michigan
  - Roseville, Michigan
  - Traverse City, Michigan
  - West Bloomfield, Michigan
  - Columbia, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Toms River, New Jersey
  - Albany, New York
  - Commack, New York
  - Kingston, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - New Bern, North Carolina
  - Salisbury, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Greensburg, Pennsylvania
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Brentwood, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Alexandria, Virginia
  - Richmond, Virginia
  - Roanoke, Virginia
  - Virginia Beach, Virginia
  - Kirkland, Washington
  - Spokane, Washington
  - Milwaukee, Wisconsin
- Austria (2):
  - Innsbruck
  - Vienna
- Roeselare, Belgium
- Canada (2):
  - London, Ontario
  - Ottawa, Ontario
- France (5):
  - Clermont-Ferrand
  - Marseille
  - Nantes
  - Pessac
  - Strasbourg
- India (8):
  - Bangalore
  - Chennai
  - Hyderabad
  - Madurai
  - Mangalore
  - Mumbai
  - Pune
  - Visakhapatnam
- Italy (3):
  - Chieti
  - Grosseto
  - Rome
- Poland (3):
  - Bydgoszcz
  - Katowice
  - Lublin
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Russia (7):
  - Kazan'
  - Kirov
  - Moscow
  - Pyatigorsk
  - Saint Petersburg
  - Samara
  - Smolensk
- Serbia (2):
  - Belgrade
  - Novi Sad
- Stockholm, Sweden
- Ukraine (5):
  - Kharkiv
  - Kiev
  - Luhansk
  - Lviv
  - Vinnitsia
- United Kingdom (5):
  - Barnsley
  - Blackburn
  - London
  - Newcastle
  - North Shields

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathis MV, Muoio BM, Andreason P, Avila AM, Farchione T, Atrakchi A, Temple RJ. The US Food and Drug Administration's Perspective on the New Antipsychotic Pimavanserin. J Clin Psychiatry. 2017 Jun;78(6):e668-e673. doi: 10.4088/JCP.16r11119. PMID 28493654
- [Derived] Ballard C, Isaacson S, Mills R, Williams H, Corbett A, Coate B, Pahwa R, Rascol O, Burn DJ. Impact of Current Antipsychotic Medications on Comparative Mortality and Adverse Events in People With Parkinson Disease Psychosis. J Am Med Dir Assoc. 2015 Oct 1;16(10):898.e1-7. doi: 10.1016/j.jamda.2015.06.021. Epub 2015 Aug 1. PMID 26239690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients were adult males or females with Parkinson's Disease Psychosis who had completed a prior double blind study with pimavanserin and were determined by the treating physician (Investigator) to benefit from continued treatment. This study did not have a fixed duration. Thus, no patients were considered to have "completed" the study.
Pre-assignment Details: Patients could be enrolled in this study as early as the final visit of the previous double-blind study, or up to 28 days following completion of the treatment period of the previous double-blind study.
Groups:
- Pimavanserin: Pimavanserin tartrate (ACP-103) tablets taken once daily by mouth for as long as the drug is considered to be tolerated and beneficial to patients
Period: Overall Study
Arm/Group | Pimavanserin
Started | 459
Completed | 0
Not Completed | 459
Not completed — Adverse Event | 88
Not completed — Death | 34
Not completed — Disease progression | 46
Not completed — Withdrawal by Subject | 167
Not completed — Physician Decision | 31
Not completed — Patient noncompliance | 25
Not completed — Lost to Follow-up | 13
Not completed — Sponsor decision | 55

BASELINE CHARACTERISTICS:
Population: Enrolled patients who received at least 1 dose of study drug
Arm/Group | Pimavanserin
Number analyzed (Participants) | 459
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176
  Male | 283
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 423
  Black/African American | 4
  Asian | 19
  Other | 13
Region of Enrollment [Number; unit: participants]
  North America | 321
  Europe | 120
  India | 18

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number (%) of Patients With Drug-related Treatment-emergent Adverse Events (AEs)
Description: Number (%) of patients with drug-related treatment-emergent AEs (i.e. AEs reported by the Investigator as possibly, probably, or highly probably related to study drug)
Time Frame: From first to last study drug dose plus 30 days
Population: Enrolled patients who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Pimavanserin
Number analyzed (Participants) | 459
Participants | 180

ADVERSE EVENTS:
Time Frame: From first to last study drug dose plus 30 days
Arm/Group | Pimavanserin
All-Cause Mortality (participants affected / at risk) | 59/459
Serious Adverse Events (participants affected / at risk) | 188/459
Other Adverse Events (participants affected / at risk) | 328/459
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=459)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 5 (5)
Cardiac arrest (Cardiac disorders) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 3 (3)
Angina pectoris (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Dyschezia (Gastrointestinal disorders) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Presbyoesophagus (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 6 (6)
Death (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Axillary pain (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 21 (23)
Urinary tract infection (Infections and infestations) | 17 (19)
Sepsis (Infections and infestations) | 7 (7)
Cellulitis (Infections and infestations) | 4 (5)
Clostridium difficile colitis (Infections and infestations) | 3 (3)
Diverticulitis (Infections and infestations) | 3 (3)
Respiratory tract infection (Infections and infestations) | 3 (3)
Bacterial sepsis (Infections and infestations) | 2 (2)
Candiduria (Infections and infestations) | 2 (2)
Coccidioidomycosis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 10 (10)
Fall (Injury, poisoning and procedural complications) | 6 (8)
Femoral neck fracture (Injury, poisoning and procedural complications) | 4 (4)
Femure fracture (Injury, poisoning and procedural complications) | 4 (5)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Nuclear magnetic resonance imaging (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 9 (9)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (4)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Parkinson's disease (Nervous system disorders) | 10 (10)
Syncope (Nervous system disorders) | 8 (9)
Dementia (Nervous system disorders) | 7 (7)
Cerebrovascular accident (Nervous system disorders) | 5 (6)
Transient ischaemic attack (Nervous system disorders) | 4 (4)
Convulsion (Nervous system disorders) | 3 (3)
Metabolic encephalopathy (Nervous system disorders) | 3 (3)
Presyncope (Nervous system disorders) | 3 (3)
Encephalopathy (Nervous system disorders) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2)
Toxic encephalopathy (Nervous system disorders) | 2 (2)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Neuroleptic malignant syndrome (Nervous system disorders) | 1 (1)
On and off phenomenon (Nervous system disorders) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Mental status change (Psychiatric disorders) | 7 (7)
Psychotic disorder (Psychiatric disorders) | 7 (7)
Hallucination (Psychiatric disorders) | 6 (6)
Hallucination, visual (Psychiatric disorders) | 2 (2)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1)
Jealous delusion (Psychiatric disorders) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renail failure (Renal and urinary disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Urinary tract obstrcution (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 11 (13)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atypical pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep brain stimulation (Surgical and medical procedures) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 5 (6)
Hypertension (Vascular disorders) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Aortic aneurysm (Vascular disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=459)
Anaemia (Blood and lymphatic system disorders) | 35 (37)
Constipation (Gastrointestinal disorders) | 46 (54)
Dysphagia (Gastrointestinal disorders) | 43 (46)
Nausea (Gastrointestinal disorders) | 39 (49)
Oedema peripheral (General disorders) | 43 (52)
Urinary tract infection (Infections and infestations) | 79 (160)
Fall (Injury, poisoning and procedural complications) | 145 (326)
Contusion (Injury, poisoning and procedural complications) | 37 (55)
Laceration (Injury, poisoning and procedural complications) | 36 (51)
Excoriation (Injury, poisoning and procedural complications) | 23 (41)
Weight decreased (Investigations) | 57 (65)
Dehydration (Metabolism and nutrition disorders) | 25 (34)
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 (42)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (38)
Dizziness (Nervous system disorders) | 43 (50)
Dementia (Nervous system disorders) | 30 (33)
Somnolence (Nervous system disorders) | 29 (33)
Parkinson's disease (Nervous system disorders) | 27 (30)
Headache (Nervous system disorders) | 23 (30)
Tremor (Nervous system disorders) | 23 (26)
Hallucination (Psychiatric disorders) | 62 (89)
Confusional state (Psychiatric disorders) | 50 (65)
Anxiety (Psychiatric disorders) | 41 (47)
Depression (Psychiatric disorders) | 39 (41)
Insomnia (Psychiatric disorders) | 34 (36)
Psychotic disorder (Psychiatric disorders) | 33 (39)
Agitation (Psychiatric disorders) | 32 (37)
Cognitive disorder (Psychiatric disorders) | 28 (33)
Orthostatic hypertension (Vascular disorders) | 40 (48)
Hypertension (Vascular disorders) | 34 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2010-07-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT00550238/Prot_000.pdf
  • Statistical Analysis Plan (2014-08-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT00550238/SAP_001.pdf